CLINICAL TRIAL: NCT03281681
Title: A Phase 1/2, Open Label, Multi-center Study of VAL-083 in Patients With Recurrent Platinum Resistant Ovarian Cancer
Brief Title: A Multi-center Study of VAL-083 in Patients With Recurrent Platinum Resistant Ovarian Cancer
Acronym: REPROVe
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Alternate study design for ovarian cancer under discussion
Sponsor: DelMar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kintara Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLM-17-001
Expanded Access: NCT03138629 (No longer available)
Record Dates: First submitted 2017-09-06; First posted 2017-09-13 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Ovarian Cancer
Keywords: adenocarcinoma of the ovary; ovarian adenocarcinoma; ovarian cancer; cancer of the ovary; ovarian neoplasm; AO; ovarian carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Dianhydrogalactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VAL-083, Dianhydrogalactitol (Experimental): VAL-083 given by intravenous infusion with a starting dose of 60 mg/m2 once weekly. If this regimen is well tolerated for at least three sequential weekly treatments the patient's dose may be escalated to 67 mg/m2 i.v. If the 67 mg/m2 dose is well tolerated for at least three sequential weekly treatments the patient's dose may be escalated to 75 mg/m2 i.v. once weekly for the remainder of the study. Dosing will be conducted once per week for a total of 16 weeks.
  Interventions: Drug: VAL-083, Dianhydrogalactitol

INTERVENTIONS:
Drug: VAL-083, Dianhydrogalactitol — VAL-083 given by intravenous infusion with a starting dose of 60 mg/m2 once weekly. If this regimen is well tolerated for at least three sequential weekly treatments the patient's dose may be escalated to 67 mg/m2 i.v. If the 67 mg/m2 dose is well tolerated for at least three sequential weekly treatments the patient's dose may be escalated to 75 mg/m2 i.v. once weekly for the remainder of the study. Dosing will be conducted once per week for a total of 16 weeks.

SUMMARY:
This is an open label, multi-center, Phase 1/2 clinical trial in subjects with recurrent adenocarcinoma of the ovary who have been previously treated with a minimum of two courses of platinum-based chemotherapy, and up to two additional cytotoxic regimens that may also have included platinum (no more than four total lines of prior therapy), with or without bevacizumab, whose cancer has recurred within six months of the most recent platinum-based chemotherapy. All eligible subjects will receive VAL 083 i.v. in a once weekly cycle until disease progression, development of other unacceptable toxicity, death, withdrawal of consent, loss to follow-up, or Sponsor ending the study, whichever occurs first.

DETAILED DESCRIPTION:
The basis of drug treatment for advanced-stage ovarian cancer in the first-line setting is platinum (cisplatin or carboplatin) plus taxane (paclitaxel or docetaxel), with or without bevacizumab. First line treatment regimens often result in high response rates, but most tumors will recur within 2 years and patients die within 3 to 4 years of diagnosis. If a patient progresses after 2 consecutive regimens without a response (refractory) or has recurrent ovarian cancer within 6 months from their last platinum-based regimen (platinum-resistant), prognosis is poor. The absence of an approved treatment or standard of care in the recurrent setting represents an unmet need.

Early NCI studies in the 1970s and 1980s support VAL-083 activity in ovarian cancer. Interest in this agent for ovarian cancer has recently re-emerged. The unique functional groups and cytotoxic mechanisms are hoped to provide a viable novel treatment option in patients with recurrent ovarian cancer that was resistant to platinum chemotherapies.

This is an open label, multi-center, Phase 1/2 clinical trial in subjects with recurrent adenocarcinoma of the ovary who have been previously treated with a minimum of two courses of platinum-based chemotherapy, and up to two additional cytotoxic regimens that may also have included platinum (no more than four total lines of prior therapy), with or without bevacizumab, whose cancer has recurred within six months of the most recent platinum-based chemotherapy.

Study subjects will initially receive VAL-083 60 mg/m2 i.v. once weekly. If this regimen is well tolerated for at least three sequential weekly treatments, the patient's dose may be escalated to 67 mg/m2 i.v. If the 67 mg/m2 dose is well tolerated for at least three sequential weekly treatments, the patient's dose may be escalated to 75 mg/m2 i.v. once weekly for the remainder of the study. Dosing will continue once weekly for 16 weeks or until disease progression, development of other unacceptable toxicity, death, withdrawal of consent, loss to follow-up, or Sponsor ending the study, whichever occurs first. The treatment plan is to enroll a minimum number of 20 subjects in Phase 1, followed by expansion of enrollment in Phase 2 using the optimal dosing regimen determined in Phase 1.

Hematological safety assessments will be conducted at Screening and weekly before each treatment. Clinical evaluations for physical examination, vital signs, disease symptoms, quality of life measures (FOSI and opioid pain medication use), adverse events and concomitant medications will be completed while the subject remains on study treatment. Radiographic assessments (computed tomography [CT] or magnetic resonance imaging [MRI]) to obtain tumor measurements and CA-125 concentration will be conducted at Screening and every 8 weeks while on study treatment, independent of dose delays and/or dose interruptions, until progression of disease is suspected.

Pharmacokinetics will be evaluated in each of the first 10 subjects who have plasma samples drawn on Day 1 of study treatment: pre-dose, then 15 ± 5 min, 30 ± 5 min, 60 ± 10 min, 120 ± 10 min, 240 ± 15 min, and 360 ± 15 min after the end of i.v. infusion with VAL-083.

A post-treatment safety assessment is to be scheduled 28 ±7 days after the last dose of study treatment.

Follow-up for subjects terminating from study for any reason other than withdrawal of consent will be done to allow an exploratory assessment of survival. All anti-tumor treatments received after discontinuing treatment with VAL-083 will be collected, if available, and survival status will also be reported to the Sponsor, on a monthly basis, when survival data are available. In addition to survival, this assessment includes outcomes for subsequent anticancer therapies including any new malignancy information. Date and cause of death will be recorded.

The primary reason for study completion and discontinuation from monthly follow-up will be captured for each study subject.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must willingly provide written consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts. (Human protection committee approval of this protocol and consent form is required).
2. Must be ≥18 years old.
3. Histologically-confirmed initial diagnosis of adenocarcinoma of the ovary (AO), excluding clear cell, low grade serous, mucinous adenocarcinoma or carcinosarcoma.
4. Subjects must have completed and failed a minimum of 2 previous lines of platinum-containing therapy (e.g., carboplatin, oxaliplatin, or cisplatin).
5. Subjects may have failed up to 2 additional cytotoxic regimens that may have included platinum.
6. Subjects must have had no more than 4 lines of prior drug therapy.
7. If treated with bevazicumab, subjects should have completed and failed treatment.
8. Subjects with BRCA mutation (positive) should have completed and failed treatment with a PARP inhibitor, or have been ineligible for treatment with a PARP inhibitor.
9. Patient must have had documented best response, disease recurrence, and date of progression based on RECIST v1.1 or CGIG criteria within 6 months from the start of last prior platinum-based therapy.
10. Formalin fixed, paraffin-embedded archival tumor available from the primary or recurrent cancer required.
11. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 and have been stable during wash-out period from prior therapy.
12. Adequate recovery from all recent surgery is required; at least 1 week must have elapsed from the time of a minor surgery; at least 21 days must have elapsed from the time of a major surgery. Must have recovered from all surgery-related toxicities to Grade 1 or less.
13. A minimum of 28 days between termination of the investigational drug and administration of VAL 083.
14. Must have recovered from all prior treatment-related toxicities to Grade 1 or less.
15. Laboratory values as follows at screening and within 3 days of planned first dose of therapy:

    1. Absolute neutrophil count (ANC) ≥ 1500/μL
    2. Hemoglobin (HgB) ≥ 9 g/dL
    3. Platelets ≥ 100,000/μL ( > 150,000/μL if prior nitrosureas)
    4. Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance > 60 mL/min (measured or calculated by the Cockcroft-Gault formula) (Cockcroft & Gault, 1976)
    5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be < 2 × ULN unless liver metastases are present, in which case they must be ≤ 5 × ULN.
    6. Total bilirubin < 1.5 × the institutional ULN, unless the patient has documented conjugated bilirubin disorder such as Gilbert's syndrome. Subjects with known Gilbert's disease who have serum bilirubin ≤ 3 × ULN (NCI CTCAE v4.03 Grade 2) may be enrolled.
    7. International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
16. Heart-rate corrected QT interval (QTc) < 450 msec on screening EKG.
17. No clinically significant cardiac conduction disorder on screening.
18. Subjects must be willing and able to comply with scheduled visits, treatment plan, and laboratory tests and be accessible for follow-up.

Exclusion Criteria:

1. Subjects with clear cell, low grade serous or mucinous adenocarcinoma, or carcinosarcoma.
2. Current history of neoplasm other than the entry diagnosis. Subjects with previous cancers treated and cured with local therapy alone may be considered with approval of the Medical Monitor.
3. Persistent Grade ≥2 toxicity from prior cancer therapy.
4. Subjects with declining ECOG performance status, defined by 1 point over a 28-day period, will be excluded.
5. Concurrent severe, intercurrent illness including, but not limited to unstable systemic disease, including ongoing or active infection, uncontrolled hypertension, serious cardiac arrhythmia requiring medication, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Any of the following cardiac conditions:

   1. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, and/or stenting up to 12 weeks before initiation of treatment with VAL-083
   2. Class III or IV heart failure as defined by the New York Heart Association functional classification system up to 6 months before initiation of treatment with VAL-083
7. Subjects with known active hepatic disease (i.e., hepatitis B or C).
8. Subjects known to be HIV positive and not on stable medication or have an AIDS-related illness.
9. Subjects with a known sensitivity to any of the products to be administered during treatment and assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Estimate Overall Response Rate | Every 8 weeks from Screening to achievement of either complete response (CR) or partial response (PR) for at least 6 months
  Overall number of tumor complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria or GCIG criteria using computed tomography (CT) or magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Safety evaluation of VAL-083 for adverse events | From Screening up to 28 days following last study treatment with VAL-083
  Using NCI CTCAE version 4 criteria to assess frequency, severity and study drug relationship of clinically significant changes in vital signs, lab test results, EKGs or any other adverse events reported while patients are receiving treatment with VAL-083
Efficacy evaluation of VAL-083 against CA-125 biomarker | From Screening to achievement of either complete response (CR) or partial response (PR) for at least 6 months
  To measure the changes in concentration of CA-125 antigen levels in blood
Progression-free Survival | Every 30 days from Screening until disease progression or patient death, whichever occurs first, for at least 6 months
  Time from start of treatment until first occurrence of progression or patient death, whichever occurs first
Comparative Progression-free Survival | Every 30 days from Screening until disease progression or patient death, whichever occurs first, for at least 6 months
  Progression-free Survival for VAL-083 compared to Progression-free Survival for patient's last treatment regimen received
Duration of Response | Every 8 weeks from Screening to achievement of either complete response (CR) or partial response (PR) for at least 6 months
  Time from start of treatment to achievement of either complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria or GCIG criteria using computed tomography (CT) or magnetic resonance imaging (MRI)
Overall Survival | Every 30 days from Screening until patient death or for at least 6 months, whichever occurs first
  Length of time from start of treatment until patient death
Cmax | Treatment Day 1 pre-dose, then 15 ± 5 min, 30 ± 5 min, 60 ± 10 min, 120 ± 10 min, 240 ± 15 min, and 360 ± 15 min after the end of the of i.v. infusion of VAL-083
  Maximum observed plasma concentration of VAL-083 in the first 10 study subjects receiving VAL-083
Tmax | Treatment Day 1 pre-dose, then 15 ± 5 min, 30 ± 5 min, 60 ± 10 min, 120 ± 10 min, 240 ± 15 min, and 360 ± 15 min after the end of the of i.v. infusion of VAL-083
  Time of maximum observed plasma concentration of VAL-083 in the first 10 study subjects receiving VAL-083
AUClast | Treatment Day 1 pre-dose, then 15 ± 5 min, 30 ± 5 min, 60 ± 10 min, 120 ± 10 min, 240 ± 15 min, and 360 ± 15 min after the end of the of i.v. infusion of VAL-083
  Area under the concentration-time curve from pre-dose (time 0) to the time of the last quantifiable concentration of VAL-083 in plasma for the first 10 study subjects receiving VAL-083
AUCinf | Treatment Day 1 pre-dose, then 15 ± 5 min, 30 ± 5 min, 60 ± 10 min, 120 ± 10 min, 240 ± 15 min, and 360 ± 15 min after the end of the of i.v. infusion of VAL-083
  Area under the concentration-time curve extrapolated to infinity for VAL-083 in plasma of the first 10 study subjects receiving VAL-083
Lambda z | Treatment Day 1 pre-dose, then 15 ± 5 min, 30 ± 5 min, 60 ± 10 min, 120 ± 10 min, 240 ± 15 min, and 360 ± 15 min after the end of the of i.v. infusion of VAL-083
  Terminal elimination rate constant determined by selection of at least 3 decreasing data points on the terminal phase of the concentration-time curve for VAL-083 in plasma of the first 10 study subjects receiving VAL-083
T 1/2 | Treatment Day 1 pre-dose, then 15 ± 5 min, 30 ± 5 min, 60 ± 10 min, 120 ± 10 min, 240 ± 15 min, and 360 ± 15 min after the end of the of i.v. infusion of VAL-083
  Terminal elimination half-life of VAL-083 in plasma of the first 10 study subjects receiving VAL-083
Quality of Life | Every 4 weeks from Screening until disease progression, for at least 6 months
  Functional Assessment of Cancer Therapy - Ovarian Symptom Index (FOSI)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J Monk, M.D., Principal Investigator — St. Joseph's Hospital and Medical Center - Phoenix, Arizona
Locations (3):
- United States (3):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Henry Ford Hospital, Detroit, Michigan
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
The Clinical Study Report for this trial will be prepared and provided to the U.S. FDA as required by applicable regulatory requirement(s). Each participating trial investigator will be provided a copy of their patient data captured in the database for this trial.